CLINICAL TRIAL: NCT02740530
Title: Improving Mobility and Cognition in Older Adults: Establishment of an Interdisciplinary Clinical Research Program Using Non-Invasive Brain Stimulation
Brief Title: Improving Mobility and Cognition in Older Adults Using Non-Invasive Brain Stimulation
Acronym: NIBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unforeseen challenges that rendered Recruitment more challenging than expected. Thus, recruitment is terminated earlier to proceed with data analysis.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Manuel Montero Odasso, MD, PhD, FRCPC, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107526
Record Dates: First submitted 2016-03-29; First posted 2016-04-15 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Executive Dysfunction; Gait Performance; Repetitive Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS Active (Experimental): High frequency pulsed repetitive magnetic stimulation at 100 % resting motor threshold will be delivered using a figure of 8 air film cooled coil attached to the Magstim® Rapid 2 machine. Resting motor threshold will be determined minimum energy needed to elicit the a reliable visible contraction in the contra-lateral first interosseous muscle using single pulse rTMS applied to the area between C1-C3 using the 10-20 international EEG electrode system. For stimulation, the coil will be positioned on the scalp corresponding to F4 then F3 electrode position using the 10-20 international EEG system. Real stimulation will consist of delivering 1200 pulses at 20 hz frequency to F4 location followed by the same stimulation to F3. The total time needed to deliver pulses is 20 minutes.
  Interventions: Device: Magstim® Rapid 2 machine
- rTMS Sham (Placebo Comparator): Sham stimulation will also involve delivering the same stimulus but with angulation of the coil at 45 degrees, which will give similar scalp sensation but unlikely to deliver magnetic stimulation to the cortex
  Interventions: Device: Magstim® Rapid 2 machine

INTERVENTIONS:
Device: Magstim® Rapid 2 machine — See Arms description
  Other Names: MAGSTIM® RAPID II SYSTEM License number 69773

SUMMARY:
This study aims to test the efficacy of a type of non-invasive brain stimulation (NIBS), known as repetitive transcranial magnetic (rTMS) stimulation, in improving mobility, particularly gait stability and variability, and executive dysfunction in older adults. The study will be conducted in forty older adults (≥60 years) with a diagnosis of executive dysfunction.

DETAILED DESCRIPTION:
The proposed study using rTMS will build upon the investigators previous work demonstrating the link between cognitive impairment, particularly executive dysfunction, and mobility/gait abnormalities in older adults, even in those labeled as "cognitively normal". Emerging evidence demonstrates that executive dysfunction is an early phenomenon in the pathway to mobility disability and subtle changes in executive function are independently associated with future falls. The investigators have piloted studies showing that pharmacological enhancement of executive function, can improve gait-motor performance and, potentially, reduce mobility decline and risk of falls. This supports the rationale for a promising intervention: enhancing cognition to prevent mobility decline and reduce risk of falls. The long-term goal is to create a clinical research program to apply rTMS as an early novel intervention for cognitive/motor interaction to ultimately delay the onset of cognitive and mobility disabilities and their devastating consequences, dementia and falls, in older adults. However, it is first necessary to study a smaller group of seniors to plan for recruitment, study retention and compliance, and to gather preliminary data as proof of principle before proceeding to a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Having executive dysfunction (defined as score below 11 out of a possible 13 in the "Montreal Cognitive Assessment -MoCA- executive score index")
* Age 60 years and older
* English speaking
* Able to ambulate 10m independently without any gait aid (eg. walker, cane)

Exclusion Criteria:

* Unable to understand or communicate in English
* Parkinsonism or any neurological disorder with residual motor deficit (eg. Major stroke, epilepsy)
* Musculoskeletal disorder detected by clinical examination which affects gait performance -Active osteoarthritis affecting lower limbs (American College of Rheumatology criteria)
* Severe depression operationalized as Geriatric Depression Scale (GDS) score>10

TMS specific exclusion criteria:

* Persons with metal anywhere in the head, excluding the mouth, including shrapnel, and screws and clips from surgical procedures
* Persons with cardiac pacemakers, implanted medication pumps, electrodes inside the heart
* Unstable heart disease
* Persons with increased intracranial pressure, as in acute large infarctions or trauma
* Previous major stroke, history seizure, Parkinson D, Huntington D.
* History of schizophrenia/schizo-affective disorder, substance use disorder within 1 year of study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Gait velocity - cm/s | Seven days

SECONDARY OUTCOMES:
Executive function, assessed as time to take to complete Trail Making A and B (TMT A and B) in seconds. | seven days

OTHER OUTCOMES:
Gait variability which is calculated as coefficient of variation (CoV) | Seven days

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Montero Odasso, MD,PhD, Principal Investigator — Lawson Health Research Institute, Western University, St. Joseph's Healthcare
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Due to the proof of principle nature of this study, our data will be crucial to establish efficacy of the intervention and furhet apply for funding for larger, clinical trial to test efectiveness

REFERENCES:
- [Background] Montero-Odasso M, Verghese J, Beauchet O, Hausdorff JM. Gait and cognition: a complementary approach to understanding brain function and the risk of falling. J Am Geriatr Soc. 2012 Nov;60(11):2127-36. doi: 10.1111/j.1532-5415.2012.04209.x. Epub 2012 Oct 30. PMID 23110433
- [Background] Montero-Odasso M, Hachinski V. Preludes to brain failure: executive dysfunction and gait disturbances. Neurol Sci. 2014 Apr;35(4):601-4. doi: 10.1007/s10072-013-1613-4. Epub 2013 Dec 24. PMID 24366243
- [Background] Shaw FE. Prevention of falls in older people with dementia. J Neural Transm (Vienna). 2007;114(10):1259-64. doi: 10.1007/s00702-007-0741-5. Epub 2007 Jun 8. PMID 17557130
- [Background] Oliver D, Connelly JB, Victor CR, Shaw FE, Whitehead A, Genc Y, Vanoli A, Martin FC, Gosney MA. Strategies to prevent falls and fractures in hospitals and care homes and effect of cognitive impairment: systematic review and meta-analyses. BMJ. 2007 Jan 13;334(7584):82. doi: 10.1136/bmj.39049.706493.55. Epub 2006 Dec 8. PMID 17158580
- [Background] Shaw FE, Bond J, Richardson DA, Dawson P, Steen IN, McKeith IG, Kenny RA. Multifactorial intervention after a fall in older people with cognitive impairment and dementia presenting to the accident and emergency department: randomised controlled trial. BMJ. 2003 Jan 11;326(7380):73. doi: 10.1136/bmj.326.7380.73. PMID 12521968
- [Background] Connolly KR, Helmer A, Cristancho MA, Cristancho P, O'Reardon JP. Effectiveness of transcranial magnetic stimulation in clinical practice post-FDA approval in the United States: results observed with the first 100 consecutive cases of depression at an academic medical center. J Clin Psychiatry. 2012 Apr;73(4):e567-73. doi: 10.4088/JCP.11m07413. PMID 22579164
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Andrews SC, Hoy KE, Enticott PG, Daskalakis ZJ, Fitzgerald PB. Improving working memory: the effect of combining cognitive activity and anodal transcranial direct current stimulation to the left dorsolateral prefrontal cortex. Brain Stimul. 2011 Apr;4(2):84-9. doi: 10.1016/j.brs.2010.06.004. Epub 2010 Jul 11. PMID 21511208
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Luber B, Kinnunen LH, Rakitin BC, Ellsasser R, Stern Y, Lisanby SH. Facilitation of performance in a working memory task with rTMS stimulation of the precuneus: frequency- and time-dependent effects. Brain Res. 2007 Jan 12;1128(1):120-9. doi: 10.1016/j.brainres.2006.10.011. Epub 2006 Nov 20. PMID 17113573
- [Background] Barr MS, Farzan F, Rajji TK, Voineskos AN, Blumberger DM, Arenovich T, Fitzgerald PB, Daskalakis ZJ. Can repetitive magnetic stimulation improve cognition in schizophrenia? Pilot data from a randomized controlled trial. Biol Psychiatry. 2013 Mar 15;73(6):510-7. doi: 10.1016/j.biopsych.2012.08.020. Epub 2012 Oct 3. PMID 23039931
- [Background] Doruk D, Gray Z, Bravo GL, Pascual-Leone A, Fregni F. Effects of tDCS on executive function in Parkinson's disease. Neurosci Lett. 2014 Oct 17;582:27-31. doi: 10.1016/j.neulet.2014.08.043. Epub 2014 Aug 30. PMID 25179996
- [Background] Reis J, Robertson EM, Krakauer JW, Rothwell J, Marshall L, Gerloff C, Wassermann EM, Pascual-Leone A, Hummel F, Celnik PA, Classen J, Floel A, Ziemann U, Paulus W, Siebner HR, Born J, Cohen LG. Consensus: Can transcranial direct current stimulation and transcranial magnetic stimulation enhance motor learning and memory formation? Brain Stimul. 2008 Oct;1(4):363-9. doi: 10.1016/j.brs.2008.08.001. Epub 2008 Oct 7. PMID 20633394
- [Background] Elder GJ, Taylor JP. Transcranial magnetic stimulation and transcranial direct current stimulation: treatments for cognitive and neuropsychiatric symptoms in the neurodegenerative dementias? Alzheimers Res Ther. 2014 Nov 10;6(9):74. doi: 10.1186/s13195-014-0074-1. eCollection 2014. PMID 25478032
- [Background] Miniussi C, Cappa SF, Cohen LG, Floel A, Fregni F, Nitsche MA, Oliveri M, Pascual-Leone A, Paulus W, Priori A, Walsh V. Efficacy of repetitive transcranial magnetic stimulation/transcranial direct current stimulation in cognitive neurorehabilitation. Brain Stimul. 2008 Oct;1(4):326-36. doi: 10.1016/j.brs.2008.07.002. Epub 2008 Oct 7. PMID 20633391
- [Background] Pascual-Leone A, Tarazona F, Keenan J, Tormos JM, Hamilton R, Catala MD. Transcranial magnetic stimulation and neuroplasticity. Neuropsychologia. 1999 Feb;37(2):207-17. doi: 10.1016/s0028-3932(98)00095-5. PMID 10080378
- [Background] Gersner R, Kravetz E, Feil J, Pell G, Zangen A. Long-term effects of repetitive transcranial magnetic stimulation on markers for neuroplasticity: differential outcomes in anesthetized and awake animals. J Neurosci. 2011 May 18;31(20):7521-6. doi: 10.1523/JNEUROSCI.6751-10.2011. PMID 21593336
- [Background] Muir SW, Gopaul K, Montero Odasso MM. The role of cognitive impairment in fall risk among older adults: a systematic review and meta-analysis. Age Ageing. 2012 May;41(3):299-308. doi: 10.1093/ageing/afs012. Epub 2012 Feb 27. PMID 22374645
- [Background] Li KZ, Roudaia E, Lussier M, Bherer L, Leroux A, McKinley PA. Benefits of cognitive dual-task training on balance performance in healthy older adults. J Gerontol A Biol Sci Med Sci. 2010 Dec;65(12):1344-52. doi: 10.1093/gerona/glq151. Epub 2010 Sep 13. PMID 20837662
- [Background] Hausdorff JM, Doniger GM, Springer S, Yogev G, Simon ES, Giladi N. A common cognitive profile in elderly fallers and in patients with Parkinson's disease: the prominence of impaired executive function and attention. Exp Aging Res. 2006 Oct-Dec;32(4):411-29. doi: 10.1080/03610730600875817. PMID 16982571
- [Background] Montero-Odasso M, Oteng-Amoako A, Speechley M, Gopaul K, Beauchet O, Annweiler C, Muir-Hunter SW. The motor signature of mild cognitive impairment: results from the gait and brain study. J Gerontol A Biol Sci Med Sci. 2014 Nov;69(11):1415-21. doi: 10.1093/gerona/glu155. Epub 2014 Sep 2. PMID 25182601
- [Background] Muir SW, Speechley M, Wells J, Borrie M, Gopaul K, Montero-Odasso M. Gait assessment in mild cognitive impairment and Alzheimer's disease: the effect of dual-task challenges across the cognitive spectrum. Gait Posture. 2012 Jan;35(1):96-100. doi: 10.1016/j.gaitpost.2011.08.014. Epub 2011 Sep 22. PMID 21940172
- [Background] Verghese J, Lipton RB, Hall CB, Kuslansky G, Katz MJ, Buschke H. Abnormality of gait as a predictor of non-Alzheimer's dementia. N Engl J Med. 2002 Nov 28;347(22):1761-8. doi: 10.1056/NEJMoa020441. PMID 12456852